CLINICAL TRIAL: NCT03858309
Title: Quantifying the Influence of Yogic Breathwork on Cerebrospinal Fluid Circulation
Brief Title: Influence of Yogic Breathwork on CSF Circulation
Acronym: CSF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Selda Yildiz, Senior Research Associate, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00019281; K99AT010158-01 (NIH)
Record Dates: First submitted 2019-02-22; First posted 2019-02-28 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: CSF Circulation
Keywords: Cerebrospinal Fluid; Cerebrospinal Fluid Flow; Cerebrospinal Fluid Circulation; Yoga; Yogic Breathwork; Magnetic Resonance Imaging; Breathing; Sleep; RT-PCMRI; CSF Flow; Slow Breathing; Respiration
MeSH Terms: conditions — Respiratory Aspiration; Hypoventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Group 1 (Experimental): Arm 1 will receive an 8-week intervention that consists of a set of breathing practices through 60-minute weekly group on-site sessions (1day/week) with a 20-minute daily home sessions (in between on-site sessions; 6 days/week).
  Interventions: Behavioral: Breathing Group 1
- Breathing Group 2 (Active Comparator): Arm 2 will receive an 8-week intervention that consists of slow breathing practices through 60-minute weekly group on-site sessions (1day/week) with a 20-minute daily home sessions (in between on-site sessions; 6 days/week).
  Interventions: Behavioral: Breathing Group 2

INTERVENTIONS:
Behavioral: Breathing Group 1 — The 8-week breathwork intervention incorporates a set of breathing practices under the guidance of a certified yoga teacher.
  Arms: Breathing Group 1
Behavioral: Breathing Group 2 — The 8-week breathwork intervention incorporates a set of slow breathing practices under the guidance of a certified yoga teacher.
  Arms: Breathing Group 2

SUMMARY:
The purpose of this research study is to determine the influence of yoga breathing practices on cerebrospinal fluid (CSF) circulation, and to find out primarily if a regular practice of 8-week yoga breathing would enhance CSF circulation as well as if the intervention would improve participant's quality of life, quality of sleep, and reduce existing stress. Participants will be randomized into two arms for different breathing practices.

DETAILED DESCRIPTION:
The purpose of this research protocol is to determine the influence of an 8-week breathing intervention on cerebrospinal fluid (CSF) circulation among healthy participants using a non-invasive real-time phase-contrast magnetic imaging (RT-PCMRI) technique. This aim will be examined by studying the changes in each participant's pre- and post-intervention CSF flow dynamics using the non-invasive RT-PCMRI technique during two MRI scans (one before and one after the 8-week intervention).

The study protocol consists of 20 healthy participants (two groups; 10 in each group with different breathing practices) undergoing an 8-week intervention, and pre-and post-intervention outcome measures.

The two 8-week interventions will be guided by two separate certified experienced yoga teachers. Both interventions will consist of 60-minute weekly group on-site sessions (1day/week) with a 20-minute daily home sessions (in between on-site sessions; 6 days/week) using home-aid practice materials. Participants' respiration data will be objectively tracked using a wearable respiration tracker device.

ELIGIBILITY:
Inclusion Criteria:

- 18-65 years of age, able to provide their consent to be in the study, available and able to participate in study activities, who can lie in supine, able to walk 15 feet, who have no prior/current mind-body practice inducing breath awareness or training such as yoga, meditation, Ta-Chi, Qi-Gong.

Exclusion Criteria:

- Inability to provide informed consent, MRI contraindications, need for muscle relaxants or anti-anxiety drugs in order to tolerate MRI, history of neurological disorders, head trauma with loss of consciousness, craniospinal disorders, spinal injury, sleep disorders, allergic or respiratory disorders, major or uncontrolled psychiatric illness or major depression, lung and heart problems, any condition requiring the use of medication that acts on the brain like stimulants, sedatives current substance abuse issues, pregnancy or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yildiz, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Breathing Group 1 | Breathing Group 2
Started (* 26 subjects were enrolled for this study for potential dropouts and to reach the target number 20 for all the study activities. * 5 subjects dropped out and/or no show up before/at their first imaging visit. * 21 subjects completed their first imaging visit, and 16 completed the study.) | 11 | 10
Completed | 9 | 7
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all 21 participants who completed enrollment and provided pre-intervention data (Active n=11, Control n=10). These participants are represented in the baseline characteristics table.
Groups:
- Total: Total of all reporting groups
Arm/Group | Breathing Group 1 | Breathing Group 2 | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.09 (14.46) | 34.00 (14.05) | 34.57 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 5 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 25.15 (4.62) | 25.89 (5.23) | 25.50 (4.81)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 126.45 (14.87) | 122.70 (21.23) | 124.67 (17.81)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.09 (11.95) | 68.60 (13.18) | 73.57 (13.16)

OUTCOME MEASURES:

1. Primary Outcome: CSF Flow Velocities
Description: We have collected cerebrospinal fluid (CSF) flow measurements during a set of breathing practices while subjects were inside the MRI scanner. MRI-based CSF flow was quantified at the level of Foramen Magnum. Data processing included the extraction of velocity waveforms of the CSF motion ( i.e, CSF velocity in cm/s) and subsequent analysis of CSF velocities across different breathing conditions. Positive CSF velocities indicate fluid motion in the cranial (upward) direction, whereas negative velocities represent fluid motion in the caudal (downward) direction.
  For the registry, descriptive statistics of CSF velocities (mean and standard deviation) are reported at pre- and post-intervention for participants completing both MRI visits with analyzable CSF data (Group 1 n=7, Group 2 n=7). No inferential statistical tests or change score analyses are included in the registry submission; all reported results are descriptive only.
Time Frame: Baseline (pre-intervention) and post-intervention (after 8 weeks).
Population: The analysis population included participants who completed both MRI visits and had analyzable CSF flow data (n=14; Group 1=7, Group 2=7). Pre- and post-intervention peak CSF velocities (maximum cranially directed and minimum caudally directed) during breathing practices were summarized in absolute units (cm/s) as mean and standard deviation.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Breathing Group 1 | Breathing Group 2
Number analyzed (Participants) | 7 | 7
cm/s
  Pre-intervention maximum (cranially directed) CSF velocity during natural breathing | 1.36 (0.27) | 1.31 (0.23)
  Post-intervention maximum (cranially directed) CSF velocity during natural breathing | 1.48 (0.42) | 1.15 (0.25)
  Pre-intervention minimum (caudally directed) CSF velocity during natural breathing | -1.92 (0.51) | -1.73 (0.41)
  Post-intervention minimum (caudally directed) CSF velocity during natural breathing | -1.68 (0.47) | -1.84 (0.45)
  Pre-intervention maximum (cranially directed) CSF velocity during slow breathing | 1.76 (0.62) | 1.48 (0.37)
  Post-intervention maximum (cranially directed) CSF velocity during slow breathing | 1.56 (0.45) | 1.35 (0.43)
  Pre-intervention minimum (caudally directed) CSF velocity during slow breathing | -2.15 (0.63) | -1.68 (0.48)
  Post-intervention minimum (caudally directed) CSF velocity during slow breathing | -1.80 (0.37) | -1.94 (0.66)
  Pre-intervention maximum (cranially directed) CSF velocity during deep abdominal breathing | 2.02 (0.64) | 1.64 (0.43)
  Post-intervention maximum (cranially directed) CSF velocity during deep abdominal breathing | 1.79 (0.57) | 1.43 (0.37)
  Pre-intervention minimum (caudally directed) CSF velocity during deep abdominal breathing | -2.12 (0.61) | -1.68 (0.47)
  Post-intervention minimum (caudally directed) CSF velocity during deep abdominal breathing | -1.90 (0.47) | -1.75 (0.55)
  Pre-intervention maximum (cranially directed) CSF velocity during deep diaphragmatic breathing | 1.88 (0.38) | 2.00 (1.31)
  Post-intervention maximum (cranially directed) CSF velocity during deep diaphragmatic breathing | 1.61 (0.58) | 1.42 (0.33)
  Pre-intervention minimum (caudally directed) CSF velocity during deep diaphragmatic breathing | -2.14 (0.61) | -2.23 (1.32)
  Post-intervention minimum (caudally directed) CSF velocity during deep diaphragmatic breathing | -1.97 (0.256) | -1.80 (0.46)
  Pre-intervention maximum (cranially directed) CSF velocity during deep chest breathing | 2.02 (0.62) | 1.49 (0.47)
  Post-intervention maximum (cranially directed) CSF velocity during deep chest breathing | 1.58 (0.45) | 1.51 (0.44)
  Pre-intervention minimum (caudally directed) CSF velocity during deep chest breathing | -2.03 (0.42) | -1.73 (0.56)
  Post-intervention minimum (caudally directed) CSF velocity during deep chest breathing | -1.74 (0.54) | -1.77 (0.53)

2. Secondary Outcome: Systolic and Diastolic Blood Pressure
Description: Systolic and diastolic blood pressure were measured participants seated at rest at pre- and post-intervention visits.
Time Frame: Baseline (pre-intervention) and post-intervention (after 8 weeks).
Population: Participants who completed both pre- and post-intervention visits and had systolic/diastolic blood pressure data collected at both time points.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Breathing Group 1 | Breathing Group 2
Number analyzed (Participants) | 9 | 7
mmHg
  Pre-intervention systolic blood pressure | 128.11 (16.07) | 117.71 (7.99)
  Post-intervention systolic blood pressure: number analyzed (Participants) | 8 | 7
  Post-intervention systolic blood pressure | 125.62 (4.55) | 118.29 (7.99)
  Pre-intervention diastolic blood pressure | 80.22 (4.08) | 66.29 (4.15)
  Post-intervention diastolic blood pressure: number analyzed (Participants) | 8 | 7
  Post-intervention diastolic blood pressure | 76.00 (3.46) | 63.43 (4.15)

3. Secondary Outcome: Body Mass Index (BMI)
Description: BMI was collected at pre- and post-intervention visits, and was calculated as weight in kilograms divided by height in meters squared (kg/m²).
Time Frame: Baseline (pre-intervention) and post-intervention (after 8 weeks).
Population: The analysis population for BMI included participants who completed both pre- and post-intervention visits and had weight and height data collected at both time points.
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | Breathing Group 1 | Breathing Group 2
Number analyzed (Participants) | 9 | 7
kg/m²
  Pre-Intervention BMI | 25.33 (1.66) | 24.33 (1.56)
  Post-Intervention BMI | 25.16 (1.57) | 24.46 (1.56)

4. Secondary Outcome: Daily Home Practice Frequency
Description: Average breathing practice frequency were measured using a wearable respiration tracker to objectively evaluate home practice throughout the intervention: frequency (days/week). Preliminary analysis estimated mean frequency (days/week) across participants. Onsite class sessions were excluded.
Time Frame: 8 weeks (daily home practice over the course of 8-week intervention).
Population: Twelve participants (6 in each group) who completed the 8-week intervention and had usable respiration tracker data. Participants without trackers or with missing data due to technical issues were excluded.
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Breathing Group 1 | Breathing Group 2
Number analyzed (Participants) | 6 | 6
days/week | 5.00 (0.82) | 5.43 (0.80)

5. Secondary Outcome: Daily Home Practice Duration
Description: Average breathing practice duration were measured using a wearable respiration tracker to objectively evaluate home practice throughout the intervention: duration (in minute). Preliminary analysis estimated mean duration (minutes) across participants. Onsite class sessions were excluded.
Time Frame: 8 weeks (daily home practice over the course of 8-week intervention).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Breathing Group 1 | Breathing Group 2
Number analyzed (Participants) | 6 | 6
minute | 21.80 (2.27) | 20.22 (0.54)

ADVERSE EVENTS:
Time Frame: 12 weeks per participant ( 2-week-pre intervention, 8-week intervention, and 2-week post-intervention).
Description: The study were to record all reportable events by study staff and through participant self-report from baseline through 2 weeks after completion of the 8-week intervention, for a total monitoring period of 12 weeks per participant (including 2-week pre-intervention, 8-week intervention, and 2-week post-intervention).
Arm/Group | Breathing Group 1 | Breathing Group 2
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
* Lack of compatible devices (iPhone or iPad) with the respiration trackers among study participants resulted in a number of participants without respiration trackers.
* Technical problems with the respiration trackers resulted in partly no data collection, or no data collection throughout the study for one subject.
* Subjects with MRI data motion artifacts and/or subjects unable to follow breathing protocol were excluded from MRI data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT03858309/Prot_SAP_000.pdf